CLINICAL TRIAL: NCT02022098
Title: A Phase I/II Randomized Study to Determine the Maximum Tolerated Dose, Safety, Pharmacokinetics and Antitumor Activity of Debio 1143 Combined With Concurrent Chemo-Radiation Therapy in Patients With Locally Advanced Squamous Cell Carcinoma of the Head and Neck.
Brief Title: Debio 1143-201 Dose-finding and Efficacy Phase I/II Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Debiopharm International SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Debio 1143-201
Record Dates: First submitted 2013-12-13; First posted 2013-12-27 (Estimated); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Cisplatin; Radiotherapy; N-benzhydryl-5-(2-(methylamino)propanamido)-3-(3-methylbutanoyl)-6-oxodecahydropyrrolo(1,2-a)(1,5)diazocine-8-carboxamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Debio 1143 (Experimental): In addition to Cisplatin and Radiotherapy, Debio 1143 in solution form will be administered orally or by feeding tube (while fasting) daily for 14 days every three weeks (on days 1-14, 22-35 and 43-56).
  Interventions: Drug: Cisplatin; Radiation: Radiotherapy; Drug: Debio 1143
- Placebo (Placebo Comparator): In addition to Cisplatin and Radiotherapy, matching placebo in solution form will be administered orally or by feeding tube (while fasting) daily for 14 days every three weeks (on days 1-14, 22-35 and 43-56).
  Interventions: Drug: Cisplatin; Radiation: Radiotherapy; Drug: Placebo

INTERVENTIONS:
Drug: Cisplatin — A total of three cycles of cisplatin will be administered in a 1-hour IV infusion on days 2, 23 and 44. Cisplatin will be administered 0.5 hours after Debio 1143.
  Other Names: Concomitant Chemotherapy
Radiation: Radiotherapy — Standard fraction radiotherapy to the primary tumour will be delivered daily for 5 days per week over 7 weeks.
  Other Names: Concomitant Radiotherapy
Drug: Debio 1143 — Debio 1143 solution
  Arms: Debio 1143
Drug: Placebo — Matching placebo solution
  Arms: Placebo

SUMMARY:
The use of multiple drugs in a single clinical trial or as a therapeutic strategy has become common, particularly in the treatment of cancer. Because traditional trials are designed to evaluate one agent at a time, the evaluation of therapies in combination requires specialized trial designs. In place of the traditional separate phase I and II trials, this trial uses a single phase I/II clinical trial to evaluate simultaneously the safety and efficacy of combination dose levels, and select the optimal combination dose.

Therefore, this is a two part trial of Debio 1143 combined with concurrent cisplatin and radiotherapy (CRT) in participants with previously untreated stage III, IVa or IVb head and neck cancer. The trial begins with an initial period of dose escalation (Phase I) to investigate the maximum tolerated dose (MTD) of Debio 1143 that can safely be given in combination with CRT.

Using the MTD determined in the Phase I portion, the randomized phase II trial in 94 participants compares Debio 1143 to placebo, both with concomitant CRT. The aim is to evaluate the efficacy and safety of Debio 1143.

ELIGIBILITY:
Inclusion Criteria:

* Meets protocol-specified criteria for qualification and contraception
* Is willing and able to comply with study procedures and restrictions related to food, drink and medications
* Voluntarily consents to participate and provides written informed consent prior to any protocol-specific procedures

Exclusion Criteria:

* Has history or current use of over-the-counter medications, dietary supplements, or drugs (including nicotine and alcohol) outside protocol-specified parameters
* Has signs, symptoms or history of any condition that, per protocol or in the opinion of the investigator, might compromise:

  1. the safety or well-being of the participant or study staff;
  2. the safety or well-being of the participant's offspring (such as through pregnancy or breast-feeding);
  3. the analysis of results

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2020-07 (Actual); Study Completion 2022-04-28 (Actual)

PRIMARY OUTCOMES:
Phase II: Percentage of participants achieving Locoregional Control (LRC) at 18 months from the end of chemo-radiation therapy (CRT) | within 4 years

SECONDARY OUTCOMES:
Phase II: Complete Response Rate (by RECIST version 1.1) at six months after completion of chemo-radiation therapy (CRT) therapy | within 5 years
Phase II: Best Overall response rate, Disease Control rate and Response Rate after 10 weeks from the end of CRT | within 5 years
Phase II: Best Overall response rate, Disease Control rate and Response Rate after 6 months from the end of CRT | within 5 years
Phase II: Locoregional control rate at 6 months and one year after completion of CRT | within 5 years
Phase II: Progression free survival rate at one year, 18 months and at 2 years as of initiation of CRT | within 5 years
Phase II: Distant relapse rate at six months, one year and 18 months after completion of CRT | within 5 years
Phase II: Disease specific survival rate one year and at 2 years as of initiation of CRT | within 5 years
Phase II: Overall survival rate at one year and at 2 years as of initiation of CRT | within 5 years
Phase II: Number of participants with clinically significant change in vital signs during participation in the trial | within 5 years
Phase II: Number of participants with Serious Adverse Events | within 5 years
Phase II: Number of participants with Adverse Events (AEs) | within 5 years
  Categories will be based on severity graded according to NCI-CTCAE version 4 criteria
Phase II: Number of participants with Laboratory Abnormalities | within 5 years
  Categories will be based on severity graded according to NCI-CTCAE version 4 criteria
Phase II: Number of participants with Late Toxicity as of initiation of CRT | within 5 years
  Categories: at 1 year, at 2 years
Phase II: Number of participants with treatment changes due to AEs | within 5 years
  Categories: Treatment discontinuation, Treatment modification

CONTACTS AND LOCATIONS:
Locations (19):
- France (17):
  - Centre Hospitalier de Bretagne Sud - HÔPITAL DU SCORFF, Lorient, BP 2233
  - C.H.U. Sud Amiens, Amiens
  - Institut Sainte-Catherine, Avignon
  - Centre Jean Perrin, Clermont-Ferrand
  - CHU Grenoble, Grenoble
  - CHD Vendée, La Roche-sur-Yon
  - Centre Guillaume le Conquérant, Le Havre
  - Centre Jean Bernard, Le Mans
  - Hôpital Nord Franche-Comté, Montbéliard
  - ICM - Val D'Aurelle, Montpellier
  - Institut Curie, Paris
  - Centre Henri Becquerel, Rouen
  - Institut de Cancérologie de l'Ouest (ICO) René Gauducheau, Saint-Herblain
  - Institut de Cancérologie Lucien Neuwirth (ICLN), Saint-Priest-en-Jarez
  - Institut Claudius Regaud, Toulouse
  - L'Institut de Cancérologie de Lorraine (ICL) Alexis Vautrin, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif
- Switzerland (2):
  - Inselspital Bern, Universitätsklinik für Radio-Onkologie, Freiburgstrasse 4, Bern
  - Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne

REFERENCES:
- [Derived] Vugmeyster Y, Ravula A, Rouits E, Diderichsen PM, Kleijn HJ, Koenig A, Wang X, Schroeder A, Goteti K, Venkatakrishnan K. Model-Informed Selection of the Recommended Phase III Dose of the Inhibitor of Apoptosis Protein Inhibitor, Xevinapant, in Combination with Cisplatin and Concurrent Radiotherapy in Patients with Locally Advanced Squamous Cell Carcinoma of the Head and Neck. Clin Pharmacol Ther. 2024 Jan;115(1):52-61. doi: 10.1002/cpt.3065. Epub 2023 Oct 23. PMID 37777832
- [Derived] Tao Y, Sun XS, Pointreau Y, Tourneau CL, Sire C, Gollmer K, Crompton P, Bourhis J. Long-term results from a clinical study of xevinapant plus chemoradiotherapy in people with high-risk locally advanced squamous cell carcinoma of the head and neck: a plain language summary. Future Oncol. 2023 Aug;19(26):1769-1776. doi: 10.2217/fon-2023-0322. Epub 2023 Jul 13. PMID 37439181
- [Derived] Tao Y, Sun XS, Pointreau Y, Le Tourneau C, Sire C, Kaminsky MC, Coutte A, Alfonsi M, Calderon B, Boisselier P, Martin L, Miroir J, Ramee JF, Delord JP, Clatot F, Rolland F, Villa J, Magne N, Elicin O, Gherga E, Nguyen F, Lafond C, Bera G, Calugaru V, Geoffrois L, Chauffert B, Damstrup L, Crompton P, Ennaji A, Gollmer K, Nauwelaerts H, Bourhis J. Extended follow-up of a phase 2 trial of xevinapant plus chemoradiotherapy in high-risk locally advanced squamous cell carcinoma of the head and neck: a randomised clinical trial. Eur J Cancer. 2023 Apr;183:24-37. doi: 10.1016/j.ejca.2022.12.015. Epub 2023 Jan 9. PMID 36796234
- [Derived] Sun XS, Tao Y, Le Tourneau C, Pointreau Y, Sire C, Kaminsky MC, Coutte A, Alfonsi M, Boisselier P, Martin L, Miroir J, Ramee JF, Delord JP, Clatot F, Rolland F, Villa J, Magne N, Elicin O, Gherga E, Nguyen F, Lafond C, Bera G, Calugaru V, Geoffrois L, Chauffert B, Zubel A, Zanna C, Brienza S, Crompton P, Rouits E, Gollmer K, Szyldergemajn S, Bourhis J. Debio 1143 and high-dose cisplatin chemoradiotherapy in high-risk locoregionally advanced squamous cell carcinoma of the head and neck: a double-blind, multicentre, randomised, phase 2 study. Lancet Oncol. 2020 Sep;21(9):1173-1187. doi: 10.1016/S1470-2045(20)30327-2. Epub 2020 Aug 3. PMID 32758455